CLINICAL TRIAL: NCT00892463
Title: Enhanced Identification of Very Early Response to Seroquel XR Added to an Antidepressant for the Treatment of Major Depressive Disorder With or Without Generalized Anxiety Disorder
Brief Title: Identifying Very Early Response to Seroquel Extended Release (XR) Augmentation for Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dr. Ayal Schaffer, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00072
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Seroquel XR; Quetiapine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Quetiapine (Seroquel) XR — 50mg/day - first 2 weeks 150mg/day - remaining 4 weeks min dose: 50mg/day max dose: 300mg/day
  Other Names: Seroquel XR

SUMMARY:
The proposed study is for a 6 week open-label clinical trial in which Seroquel XR is added to a selective serotonin reuptake inhibitor (SSRI) medication for the treatment of depressive and/or anxiety symptoms. Each subject will self-report changes in symptoms, functional impairment, etc. on a twice daily basis using a handheld computer (HHC) that transmits real-time symptoms reports to a central database. Each subject will be assessed in-person on a weekly or biweekly basis during the course of the study.

DETAILED DESCRIPTION:
This study is a 6-week open-label clinical trial in which Seroquel XR is added to an antidepressant medication for the treatment of MDD with or without comorbid generalized anxiety disorder. Patients who are currently experiencing a depressive episode that has not responded to an adequate trial of an antidepressant will be eligible to participate. During the course of augmentation treatment with Seroquel XR, each subject will regularly enter information on symptom severity and functional impairment into their handheld computer, and this information will be wirelessly transmitted to a central database.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of major depressive disorder, currently depressed with or without a comorbid generalized anxiety disorder as determined by DSM-IV diagnostic criteria (confirmed using the MINI)
2. Outpatient status
3. 17-item Hamilton Depression Rating Scale (HAM-D) score of ≥ 18
4. Treatment with any of the following antidepressant medications for the past 4 weeks at a minimum therapeutic dose

Exclusion Criteria:

1. Diagnosis of a past or current bipolar disorder
2. Current psychotic symptoms
3. Substance-induced mood disorder
4. Substance or alcohol dependence
5. Prominent current suicidal ideation as defined by a HAM-D item 3 (suicide item) score of ≥ 3
6. Current treatment with more than one antidepressant medication
7. Current treatment with an tricyclic (TCA) antidepressant or monoamine oxidase inhibitor (MAOI)
8. A patient with Diabetes Mellitus (DM)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The QIDS-SR16 (Quick Inventory of Depressive Symptomatology - Self-report) | Once Daily for 6 weeks

SECONDARY OUTCOMES:
HADS (Hamilton Anxiety Depression Scale) VADIS | Once/twice Daily for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ayal Schaffer, MD, Principal Investigator — Sunnybrook Health Sciences Centre - University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada